CLINICAL TRIAL: NCT00459186
Title: A Phase I/II Study of RAD001 With Docetaxel in the Treatment of Metastatic, Androgen Independent Prostate Cancer
Brief Title: The Use of RAD001 With Docetaxel in the Treatment of Metastatic, Androgen Independent Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Mary-Ellen Taplin, MD, Associate Professor of Medicine, HMS, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-184
Record Dates: First submitted 2006-01-23; First posted 2007-04-11 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Metastatic, Androgen Independent Prostate Cancer; Prostate Cancer
Keywords: prostate cancer; RAD001; mTOR inhibition; docetaxel
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Everolimus; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 Followed by RAD001 + Docetaxel (Experimental): RAD001 10 mg daily for 2 weeks, followed by RAD001 + Docetaxel at one of three doses: 5 mg RAD001 and docetaxel at 60 mg/m2, 10 mg RAD001 and docetaxel at 60 mg/m2, and 10 mg RAD001 and docetaxel at 70 mg/m2. RAD001 was given daily. Docetaxel was given every 3 weeks by intravenous infusion. Patients also received prednisone 5 mg by mouth twice daily.
  Interventions: Drug: RAD001; Drug: Docetaxel; Drug: Prednisone

INTERVENTIONS:
Drug: RAD001 — Daily for two weeks
Drug: Docetaxel — Infusion once per cycle
Drug: Prednisone — Prednisone 5 mg by mouth twice daily

SUMMARY:
The purpose of this study is to evaluate the safety and optimal dose of RAD001 and docetaxel plus prednisone in men with hormone refractory, metastatic prostate cancer (Phase I).

Once an appropriate dose is reached, the purpose then will be to determine the response rate of docetaxel plus RAD001 (Phase II).

DETAILED DESCRIPTION:
* Patients will be designated into one of two groups based upon the results of a FDG-PET scan.
* A patient with a baseline positive scan will have serum drawn for baseline serum proteomics assessment then be treated with RAD001 daily for two weeks. On day 10-14, another FDG-PET scan and serum assessment will be performed. An optional bone marrow biopsy may also be done. On day 15, patients will enter the Phase I portion of the trial at the current enrolling dosage or if Phase I is completed patients will enter Phase II.
* A patient that does not have a positive scan will enter directly into the Phase I trial or Phase II depending on which trial is currently enrolling.
* Phase I trial patients will have weekly laboratory evaluations and clinical evaluation every three weeks.
* Phase II trial patients will have laboratory evaluations on day one and day eight and clinical evaluation every three weeks.
* The maximum duration of the trial is one year of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate with radiographic evidence of metastatic disease.
* Willingness to undergo a baseline tumor biopsy.
* Castrate levels of testosterone (testosterone < 50 ng/dL) on androgen deprivation therapy (ADT) with evidence of progression on ADT. GnRH therapy will be continued for those on it at baseline
* Patient must have suspected tumor in an area that is safe to biopsy.
* Other prior hormonal interventions or experimental approaches are allowed. These therapies must have been discontinued for a minimum of 28 days with cancer progression.
* Prior or concurrent use of bisphosphonates is allowed.
* One prior non-taxane chemotherapy allowed
* ≥ 3 weeks since major surgery; ≥ 4 weeks since radiotherapy; ≥ 8 weeks since prior strontium-89 or samarium 153
* Performance Status: ECOG 0 or 1
* ANC > 1,500/_l; platelets > 100,000/_l; total Bilirubin < upper limit of normal; AST and ALT < 3 x upper limits of normal; creatinine < 1.5 x upper limits of normal; total fasting cholesterol < 350 mg/dl; total triglycerides < 300 mg/dl

Exclusion Criteria:

* Ongoing oral steroid use. Patients with a history of oral steroid use are eligible as long as the steroids have been discontinued prior to study entry. Ongoing topical and/or inhaled steroid use is allowed.
* Prior taxane chemotherapy
* Prior mTOR inhibitors (RAD001, rapamycin, CCI-779)
* Currently active second malignancy other than non-melanoma skin cancer.
* Ongoing peripheral neuropathy of Grade 2

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Oregon Health Science University, Portland, Oregon

REFERENCES:
- [Derived] Courtney KD, Manola JB, Elfiky AA, Ross R, Oh WK, Yap JT, Van den Abbeele AD, Ryan CW, Beer TM, Loda M, Priolo C, Kantoff P, Taplin ME. A phase I study of everolimus and docetaxel in patients with castration-resistant prostate cancer. Clin Genitourin Cancer. 2015 Apr;13(2):113-23. doi: 10.1016/j.clgc.2014.08.007. Epub 2014 Oct 22. PMID 25450031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Genitourinary Oncology clinics of Dana-Farber Cancer Institute and the Knight Cancer Institute at Oregon Health and Science University between November, 2005 and October, 2008
Period: Single Agent RAD001
Arm/Group | RAD001 Followed by RAD001 + Docetaxel
Started | 19
Completed | 18
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: PET Imaging and Assessment
Arm/Group | RAD001 Followed by RAD001 + Docetaxel
Started | 18
Completed | 15
Not Completed | 3
Not completed — Adverse Event | 3
Period: Combination RAD001 + Docetaxel
Arm/Group | RAD001 Followed by RAD001 + Docetaxel
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Number of baseline participants represents the number who received at least one dose of investigational agent (did not withdraw before treatment).
Arm/Group | RAD001 Followed by RAD001 + Docetaxel
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 62 [50 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Free of Dose Limiting Toxicity
Description: A dose limiting toxicity was defined as an adverse event or laboratory abnormality that occurs to patients on the Phase I portion of the trial, during the first 21 days following the first dose of RAD001/docetaxel during cycle 1, judged to be related to RAD001/docetaxel and meeting any of the following criteria:
  Hematologic Toxicity:
  CTCAE grade 4 neutropenia > 7 days or any Grade 3 or 4 neutropenia with fever Or CTCAE grade 3 or 4 thrombocytopenia > 7 days
  Non-hematologic toxicity:
  The occurrence of non-hematologic CTCAE grade 3 or 4 adverse events will be considered dose limiting, except for the following:
  1. CTCAE grade 3 nausea or grade 3 or 4 vomiting CTCAE grade 3 or 4 vomiting will only be considered dose limiting if it occurs despite the use of standard anti-emetics.
  2. CTCAE grade 3 or 4 fever identified with a source (i.e. infection, tumor)
  3. CTCAE grade 3 or 4 alkaline phosphatase.
Time Frame: 21 days
Population: Patients who received combination treatment with RAD001 + Docetaxel
Measure: Number; unit: participants
Arm/Group | RAD001 Followed by RAD001 + Docetaxel
Number analyzed (Participants) | 15
participants | 14

2. Secondary Outcome: Response Based on PET Scan
Description: Patients were scanned using Positron Emission Tomography (PET) before and after receiving single agent RAD001. Patients were classified as having partial metabolic response, stable metabolic disease, or progressive metabolic disease based on changes in PET imaging from baseline to post-treatment. A positive FDG-PET for the purposes of this study consisted of a visualized area of abnormal increased FDG uptake that matched the anatomic location of an abnormality seen on bone scan or CT. Metabolic response was assessed for percent change in SUVmax according to the criteria of the European Organization for Research and Treatment of Cancer (EORTC) : partial metabolic response (PMR) ≤ -25%; stable metabolic disease (SMD) -25% + 25%; progressive metabolic disease (PMD) > 25%.
Time Frame: 10 to 14 days after study entry
Population: All patients receiving at least one dose of RAD001
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | RAD001 Followed by RAD001 + Docetaxel
Number analyzed (Participants) | 18
percentage of participants
  Partial Metabolic Response | 22 [8 to 44]
  Stable Metabolic Disease | 67 [45 to 84]
  Progressive Metabolic Disease | 11 [2 to 31]

ADVERSE EVENTS:
Arm/Group | RAD001 Followed by RAD001 + Docetaxel
Serious Adverse Events (participants affected / at risk) | 13/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 Followed by RAD001 + Docetaxel (N=18)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Cholecystitis (Hepatobiliary disorders) | 1
Infection with Grade 3-4 neutrophils - lung (Infections and infestations) | 1
Infection with Grade 0-2 neutrophils - lung (Infections and infestations) | 1
Leukopenia (Investigations) | 6
Neutropenia (Investigations) | 8
Thrombocytopenia (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 Followed by RAD001 + Docetaxel (N=18)
Constipation (Gastrointestinal disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 8
Hemorrhoids (Gastrointestinal disorders) | 1
Muco/stomatitis by exam - oral cavity (Gastrointestinal disorders) | 4
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
GI-other (Gastrointestinal disorders) | 1
Abdomen - pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 8
Fever w/o neutropenia (General disorders) | 2
Rigors/chills (General disorders) | 1
Edema limb (General disorders) | 2
Infection with Grade 0-2 neutrophils - upper airway (Infections and infestations) | 2
Weight loss (Investigations) | 1
Elevated AST/SGOT (Investigations) | 4
Hypercholesterolemia (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Extremity-limb - pain (Musculoskeletal and connective tissue disorders) | 1
Joint - pain (Musculoskeletal and connective tissue disorders) | 1
Muscle - pain (Musculoskeletal and connective tissue disorders) | 1
Taste disturbance (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Nose - hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
Throat/pharynx/larynx - pain (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Nail changes (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No